CLINICAL TRIAL: NCT02218502
Title: Regional Study Into the Performance and Cost-effectiveness of Simple Ultrasound-based Rules Compared to the Currently Used Risk of Malignancy Index in the Diagnosis of Ovarian Cancer
Brief Title: Study Into a New Diagnostic Tool (Simple Ultrasound-based Rules) in Patients With Adnexal Masses
Acronym: SUBSONiC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: interim analysis showed incorrect use of simple rules
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Laurentius Hospital Roermond (Unknown); St.Jans Gasthuis Weert (Unknown); VieCuri Medical Centre (Other); Orbis Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: NL44181.068.13
Record Dates: First submitted 2014-07-07; First posted 2014-08-18 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Ovarian Carcinoma; Ovarian Cancer; Ovarian Mass; Ovarian Cyst
Keywords: Ovarian cancer; Diagnosis; Risk of Malignancy Index; RMI; Ultrasound; Simple ultrasound-based rules; DW-MRI; Subjective assessment
MeSH Terms: conditions — Ovarian Neoplasms; Ovarian Cysts; Disease

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- If simple rules are conclusive (Other): All patients included will undergo an ultrasound scan in which both the RMI and simple ultrasound-based rules are applied. This scan will take place in the hospital of inclusion. For 80% of all patients, this will be the only intervention.
  Interventions: Other: Ultrasound by general gynaecologist
- If simple rules are inconclusive (Other): If the simple ultrasound-based rules, used in the first ultrasound scan, yield an inconclusive result (approx. 20% of all patients), patients are refered to the center hospital to undergo a second ultrasound (by an expert) and a DW-MRI scan. Furthermore, these group of patients will be asked to give an extra blood sample in order to perform translational research and validate new biomarkers in the diagnosis of ovarian cancer.
  Interventions: Other: Ultrasound by general gynaecologist; Other: Ultrasound by an expert ultrasonographist; Other: DW-MRI; Other: Give blood sample

INTERVENTIONS:
Other: Ultrasound by general gynaecologist — All patients will undergo an ultrasound by a general gynaecologist at the moment of inclusion. Based on this ultrasound, the gynaecologist will use both the RMI and the simple rules to predict the chance of malignancy.
Other: Ultrasound by an expert ultrasonographist — Patients in which the simple rules yield an inconclusive result (about 20% of all patients) will undergo a second ultrasound scan. This scan is performed by an expert in gynaecological ultrasound.
  Arms: If simple rules are inconclusive
Other: DW-MRI — Patients in which the simple rules yield an inconclusive result (about 20% of all patients) will undergo a diffusion weighted MRI.
  Arms: If simple rules are inconclusive
Other: Give blood sample — Patients in which the simple rules yield an inconclusive result (about 20% of the patients) will be asked for an extra blood sample. We will use these materials to perform translational research and validate new biomarkers in the diagnosis of ovarian cancer.
  Arms: If simple rules are inconclusive

SUMMARY:
This study is performed to compare the diagnostic performance and cost-effectiveness of different diagnostic methods for differentiating benign from malignant adnexal (ovary or Fallopian tube) masses: the Risk of Malignancy Index (RMI) will be compared with a two-step triage test called "simple ultrasound-based rules" supplemented -if necessary- with either subjective assessment by an expert sonographer or Diffusion Weighted - Magnetic Resonance Imaging (DW-MRI). The investigators will test the hypothesis that this two-step triage test will have better diagnostic accuracy than the RMI and therefore will improve the management of women with adnexal masses.

DETAILED DESCRIPTION:
Estimating whether an adnexal mass is malignant or not is essential in the preoperative management of adnexal masses. Recognizing cancer means treatment is not delayed and appropriate staging or debulking surgery can be carried out after referral to specialized surgical centers. Vice versa, benign lesions may be managed conservatively or with minimal invasive surgery in non-centre hospitals. This will limit morbidity and will avoid unnecessary costs: laparoscopic surgery offers lower estimated blood loss, shorter hospital stay, and fewer postoperative complications with an improved quality of life and faster return to normal functioning.

There are several methods to distinguish benign from malignant adnexal masses. The commonly used method in clinical practice is the Risk of Malignancy Index (RMI). The RMI is an easy to use scoring system recommended by many national guidelines concerning the management of ovarian masses, including the national guideline in the Netherlands. The RMI combines ultrasound variables, menopausal status and serum CA125 into a score used to predict the risk of ovarian cancer before surgery. However, the reported sensitivity and specificity of RMI at a cut-off value of 200 are relatively low; 75-80% and 85-90%, respectively.

Another method called 'simple ultrasound-based rules' (simple rules), uses different morphological ultrasound features of adnexal masses (without including menopausal status or serum CA125 measurement). It includes five simple ultrasound-based rules to predict malignancy (M-rules) and five rules to predict a benign tumor (B-rules). If both or none of the M- and B-rules are met (20% of the patients) the test is inconclusive. Recent reports show that simple rules might be superior to the RMI. In adnexal masses for which the simple ultrasound rules yield an inconclusive result, subjective assessment of Gray-scale and color Doppler ultrasound images by an experienced ultrasound examiner can be used as a second stage test to achieve an optimal diagnostic performance. Subjective assessment by an expert sonographer is superior to any scoring system or mathematical model when classifying adnexal masses as benign or malignant. However, it is not feasible and efficient that every patient would undergo an expert ultrasonography. Therefore, this method is better used as a second stage test.

Another option is to use Diffusion Weighted - Magnetic Resonance Imaging (DW-MRI) as a second stage test, when the simple rules yield an inconclusive result. The use of MRI - when interpret by specialized radiologists- also seems to be superior to RMI in the preoperative identification of adnexal masses.

The Risk of Malignancy Index (RMI) is the current standard in differentiating benign from malignant adnexal masses. The simple ultrasound-based rules as a first stage triage test followed by either subjective assessment by an experienced ultrasound examiner or DW-MRI in case the simple rules are inconclusive, is the test of comparison. Both the RMI and the simple rules will be performed in the regional hospitals and MUMC+ by general gynaecologists during the same ultrasound scan. Only when the simple rules are inconclusive the patient will be referred to the MUMC+ for a second stage test. From previous publications it can be deducted that this will be in approximately 20% of patients. Approximately 80% of patients will not need any additional second stage test.

The histology of the surgically removed adnexal masses is the clinical reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Female patient;
* Diagnosed in one of the participating centers with at least one pelvic mass that is suspected to be of ovarian origin;
* Are to undergo surgery in order to obtain a final histological diagnosis;
* 18 years of age or older.

Exclusion Criteria:

* Pregnant patients;
* Patients aged under 18 years;
* Patients in whom the surgery does not take place, or takes place more than 120 days after RMI and simple ultrasound-based rules are performed;
* Patients with a prior bilateral oophorectomy;
* Patients with insufficient or missing data;
* Patients who do not give or are incapable of giving an informed consent;
* Patients who are not able or willing to travel to the center hospital for additional diagnostic procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-10-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity | This analysis will take place after completing the inclusion of patients (approx. 2 years)
  Sensitivity is defined as the percentage of women with ovarian cancer diagnosed with a malignancy by respectively the RMI and the two-step test. Specificity is defined as the percentage of correctly diagnosed benign masses.
Likelihood ratios | This analysis will take place after completing the inclusion of patients (approx. 2 years)
  The positive likelihood ratio is calculated by dividing the sensitivity by 100 minus the specificity. The negative likelihood ratio is calculated as the sensitivity minus 100 divided by the specificity.
positive and negative predictive values | This analysis will take place after completing the inclusion of patients (approx. 2 years)
  The positive predictive value is defined as the percentage of patients with a positive test result by respectively RMI and simple rules having malignant disease. The negative predictive value is defined as the percentage of patients with a negative test result having benign disease.
cost-effectiveness | This analysis will take place after completing the inclusion of patients (approx. 2 years)
  The economic evaluation will explore the potential cost-effectiveness of RMI versus the triage test. Incremental cost-effectiveness will be expressed as the costs per correct diagnosis (i.e. either true positive or false negative for malignancy based on histology) including the costs of surgical management following diagnosis. The analysis will take a hospital perspective including all costs from inclusion up to hospital discharge following surgery. As not all data necessary for comparison between the diagnostic strategies will be collected empirically and surgical management will be based on RMI, a simple decision analytic model will be constructed. The comparative sensitivity, specificity and costs of the diagnostic strategies including surgical management for the diagnostic work up of patients with at least one pelvic mass that is suspected to be of ovarian origin, will explicitly be incorporated in the model.
Budget Impact Analysis (BIA) | This analysis will take place after completing the inclusion of patients (approx. 2 years)
  A budget impact analysis will be performed according to the ISPOR guidelines. The BIA addresses the financial stream of consequences related to the uptake and diffusion of the triage test to assess affordability. The budget impact will depend on both the costs of the diagnostic strategies, the effect in terms of correct diagnosis, as well as potential future levels of uptake of the triage test. All these elements which determine the potential budget impact will be addressed in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Evelyne MJ Meys, LLM, BsC, Study Director — Maastricht University Medical Center; Toon van Gorp, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (5):
- Netherlands (5):
  - Maastricht University Medical Centre (MUMC+), Maastricht
  - Laurentius Ziekenhuis Roermond, Roermond
  - Orbis Medical Sittard, Sittard
  - VieCuri Venlo, Venlo
  - St.Jans Gasthuis Weert, Weert

REFERENCES:
- [Background] Weber S, McCann CK, Boruta DM, Schorge JO, Growdon WB. Laparoscopic surgical staging of early ovarian cancer. Rev Obstet Gynecol. 2011;4(3-4):117-22. PMID 22229064
- [Background] Timmerman D, Ameye L, Fischerova D, Epstein E, Melis GB, Guerriero S, Van Holsbeke C, Savelli L, Fruscio R, Lissoni AA, Testa AC, Veldman J, Vergote I, Van Huffel S, Bourne T, Valentin L. Simple ultrasound rules to distinguish between benign and malignant adnexal masses before surgery: prospective validation by IOTA group. BMJ. 2010 Dec 14;341:c6839. doi: 10.1136/bmj.c6839. PMID 21156740
- [Background] Timmerman D, Testa AC, Bourne T, Ameye L, Jurkovic D, Van Holsbeke C, Paladini D, Van Calster B, Vergote I, Van Huffel S, Valentin L. Simple ultrasound-based rules for the diagnosis of ovarian cancer. Ultrasound Obstet Gynecol. 2008 Jun;31(6):681-90. doi: 10.1002/uog.5365. PMID 18504770
- [Background] Van Gorp T, Veldman J, Van Calster B, Cadron I, Leunen K, Amant F, Timmerman D, Vergote I. Subjective assessment by ultrasound is superior to the risk of malignancy index (RMI) or the risk of ovarian malignancy algorithm (ROMA) in discriminating benign from malignant adnexal masses. Eur J Cancer. 2012 Jul;48(11):1649-56. doi: 10.1016/j.ejca.2011.12.003. Epub 2012 Jan 5. PMID 22226481
- [Background] Valentin L, Jurkovic D, Van Calster B, Testa A, Van Holsbeke C, Bourne T, Vergote I, Van Huffel S, Timmerman D. Adding a single CA 125 measurement to ultrasound imaging performed by an experienced examiner does not improve preoperative discrimination between benign and malignant adnexal masses. Ultrasound Obstet Gynecol. 2009 Sep;34(3):345-54. doi: 10.1002/uog.6415. PMID 19585547
- [Background] Dodge JE, Covens AL, Lacchetti C, Elit LM, Le T, Devries-Aboud M, Fung-Kee-Fung M; Gynecology Cancer Disease Site Group. Preoperative identification of a suspicious adnexal mass: a systematic review and meta-analysis. Gynecol Oncol. 2012 Jul;126(1):157-66. doi: 10.1016/j.ygyno.2012.03.048. Epub 2012 Apr 6. PMID 22484399
- [Background] Tingulstad S, Hagen B, Skjeldestad FE, Halvorsen T, Nustad K, Onsrud M. The risk-of-malignancy index to evaluate potential ovarian cancers in local hospitals. Obstet Gynecol. 1999 Mar;93(3):448-52. PMID 10074998
- [Background] Tingulstad S, Hagen B, Skjeldestad FE, Onsrud M, Kiserud T, Halvorsen T, Nustad K. Evaluation of a risk of malignancy index based on serum CA125, ultrasound findings and menopausal status in the pre-operative diagnosis of pelvic masses. Br J Obstet Gynaecol. 1996 Aug;103(8):826-31. doi: 10.1111/j.1471-0528.1996.tb09882.x. PMID 8760716
- [Background] Jacobs I, Oram D, Fairbanks J, Turner J, Frost C, Grudzinskas JG. A risk of malignancy index incorporating CA 125, ultrasound and menopausal status for the accurate preoperative diagnosis of ovarian cancer. Br J Obstet Gynaecol. 1990 Oct;97(10):922-9. doi: 10.1111/j.1471-0528.1990.tb02448.x. PMID 2223684
- [Background] Mauskopf JA, Sullivan SD, Annemans L, Caro J, Mullins CD, Nuijten M, Orlewska E, Watkins J, Trueman P. Principles of good practice for budget impact analysis: report of the ISPOR Task Force on good research practices--budget impact analysis. Value Health. 2007 Sep-Oct;10(5):336-47. doi: 10.1111/j.1524-4733.2007.00187.x. PMID 17888098
- [Derived] Meys EM, Rutten IJ, Kruitwagen RF, Slangen BF, Bergmans MG, Mertens HJ, Nolting E, Boskamp D, Beets-Tan RG, van Gorp T. Investigating the performance and cost-effectiveness of the simple ultrasound-based rules compared to the risk of malignancy index in the diagnosis of ovarian cancer (SUBSONiC-study): protocol of a prospective multicenter cohort study in the Netherlands. BMC Cancer. 2015 Jun 26;15:482. doi: 10.1186/s12885-015-1319-5. PMID 26111920